CLINICAL TRIAL: NCT07345650
Title: Dynamic Compliance-Guided Personalized PEEP During Laparoscopic Bariatric Surgery: Effects on Intraoperative Respiratory Parameters
Status: Active, not recruiting | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KAEK-21/1045
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Obesity (Body Mass Index >30 kg/m2); Atelectasis, Postoperative; PEEP With Dynamic Compliance; Individualized PEEP
Keywords: obesity; bariatric surgery; postoperative atelectasis; individualized peep
MeSH Terms: conditions — Obesity; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — arterial blood gas
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SP-standard peep: individuals monitored by standard PEEP
- KP-individualized peep: individuals monitored by individualized PEEP
  Interventions: Device: Individualized approach

INTERVENTIONS:
Device: Individualized approach — individuals were compared by using of a personalized peep or not
  Groups: KP-individualized peep

SUMMARY:
Atelectasis may be encountered in the patient population aged 18-65 years undergoing elective laparoscopic bariatric surgery under general anesthesia with endotracheal intubation. The aim of this study is to compare oxygenation, postoperative atelectasis, and postoperative respiratory complications between the fixed PEEP application (SP Group) and personalized PEEP application (KP Group). In the SP Group, ventilation will be applied with PEEP = 8 cmH2O, tidal volume = 8 ml/kg, and respiratory rate to maintain EtCO2 between 35-40, and this ventilation mode was maintained throughout the entire surgery. In the KP Group, ventilation was applied with tidal volume = 8 ml/kg, PEEP = 4 cmH2O, and respiratory rate to maintain EtCO2 between 35 -40, and dynamic compliance was noted 1 minute after the onset of pneumoperitoneum at 12 mmHg. Subsequently, the PEEP value wastitrated every 2 minutes by increasing it by 2 cmH2O until the level providing the highest dynamic compliance value is reached. If the dynamic compliance value does not increase in two consecutive measurements, the previous PEEP value was defined as the patient's "personalized PEEP" value, and ventilation was continued with this PEEP value until the end of the surgery. In all patients, arterial blood gas (ABG) was obtained 10 minutes after anesthesia induction, at the 10th and 30th minutes of pneumoperitoneum, and 10 minutes after pneumoperitoneum is terminated.Patients were transferred to the recovery room after anesthesia is discontinued, and arterial blood gas sampling and lung ultrasound was performed at 30 minutes postoperatively.

On postoperative day 1, presence of atelectasis was assessed with lung ultrasound, and SpO2 was recorded at 4th, 12th, and 24th hours postoperatively. Within 4 hours postoperatively, patients in need of supplemental oxygen were recorded(SpO2 92% was decided as cut-off value). After the 4th hour, the number of patients requiring supplemental oxygen after the 4th hour was recorded and compared in both groups. Data were collected and recorded using a standardized paper-based data collection form. A power analysis measurement (post-hoc test) is planned to be performed. If the power analysis exceeds 80% between the groups, the study will be terminated. Data collection was completed after reaching the planned number of volunteers. The study results will be evaluated using the SPSS statistical analysis program. Numerical data between groups (SP vs. KP) will be evaluated using the ANOVA test or Kruskal Wallis test, while categorical data will be evaluated using the chi-square test or Fisher exact test. P<0.05 will be considered statistically significant, and univariate and multivariate analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

Adult women and men aged 18 to 65 years Scheduled for elective laparoscopic bariatric surgery American Society of Anesthesiologists (ASA) physical status I-III Body mass index (BMI) > 30 kg/m² Provision of written informed consent

Exclusion Criteria:

Age < 18 years or > 65 years Not scheduled for bariatric surgery ASA physical status IV-V Body mass index (BMI) < 30 kg/m² Refusal or inability to provide inHistory of Chronic Obstructive Pulmonary Disease (GOLD III and IV) History of severe/uncontrolled bronchial asthma Severe restrictive lung disease History of pulmonary metastases History of thoracic surgery Requiring preoperative thoracic drainage Requiring preoperative renal replacement therapy Congestive heart failure (NYHA Class III and IV)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult women and men aged 18 to 65 years who were scheduled for elective laparoscopic bariatric surgery. Eligible participants had an American Society of Anesthesiologists (ASA) physical status of I-III and a body mass index (BMI) greater than 30 kg/m². All participants provided written informed consent prior to enrollment.
  Patients were excluded if they were younger than 18 years or older than 65 years, were not scheduled for bariatric surgery, had an ASA physical status of IV-V, or a BMI less than 30 kg/m². Additional exclusion criteria included refusal or inability to provide informed consent; a history of chronic obstructive pulmonary disease (COPD) classified as GOLD stage III or IV; severe or uncontrolled bronchial asthma; severe restrictive lung disease; a history of pulmonary metastases or previous thoracic surgery; the requirement for preoperative thoracic drainage; the need for preoperative renal replacement therapy; and congestive heart fail
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
LUSS score (lung ultrasound severity score) | 6 months
  Lung aeration was assessed using the Lung Ultrasound Score (LUS). Each lung was divided into six regions (anterior, lateral, and posterior areas, each subdivided into upper and lower regions), resulting in a total of 12 regions. Each region was scored from 0 to 3 based on ultrasound findings, with higher scores indicating greater loss of lung aeration. The total LUS ranged from 0 to 36.
compliance in individualized and non-individualized peep group | 6 months
  Compliance was assessed intraoperatively in both the individualized PEEP group and the non-individualized (fixed PEEP) group.In the individualized PEEP group, PEEP was titrated based on dynamic compliance, and respiratory system compliance was recorded at the PEEP level that yielded the highest dynamic compliance value for each patient.In the non-individualized PEEP group, a predefined fixed PEEP level was applied throughout the procedure, and respiratory system compliance was measured at this fixed PEEP level.
arterial blood gas analysis | 6 months
  Arterial blood gas analysis was performed to assess arterial oxygenation. The partial pressure of arterial oxygen (PaO₂) was recorded at predefined intraoperative time points and analyzed to determine significant differences between the individualized PEEP and fixed PEEP groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study is not over yet, this is the reason why IPD might not be shared yet.